CLINICAL TRIAL: NCT01644409
Title: Urgent-SQ Implant in Treatment of Overactive Bladder Syndrome: Nine-year Follow-up Study
Brief Title: Urgent-SQ in Treatment of Overactive Bladder Syndrome: 9-yr Follow up
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Dick Janssen, MD researcher, Radboud University Medical Center
Other Study IDs: USQ-9yr; USQ-9yr (Other: Radboud University Nijmegen Medical Centre)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Overactive Bladder; Urinary Frequency or Urgency Adverse Event; Urinary Incontinence, Urge
Keywords: OAB; Overactive bladder; Urgency; Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Long term open label study on safety and durability of the Urgent-SQ tibial implant device for refractory overactive bladder syndrome (OAB).

DETAILED DESCRIPTION:
This is a follow-up study of the study by van der Pal et al. (see reference). The Urgent-SQ is an ankle (tibail) implant that is used for on demand electical stimulation that stimulates the tibial nerve for the treatment of overactive bladder syndrome (OAB). The implant is placed via an minimal invasive surgical procedure. The implant can be activated with an external pulse generator.

This study by van de Pal et al. was conducted with the approval of the local Medical Ethical Committee and with a one year systematic follow-up of eight patients. Since then, follow-up up and use of the device was open-label.

This study reports on the long-term (9yrs) the safety and durability of the Urgent-SQ implant in these eight patients.

Parameters evaluated were local pain and discomford at the site of the implant, AE's related to the implant or the use of the implant. Current use of the treatment and effectivity of the treatment.

van der Pal F, van Balken MR, Heesakkers JP, Debruyne FM, Bemelmans BL.Implant-Driven Tibial Nerve Stimulation in the Treatment of Refractory Overactive Bladder Syndrome: 12-Month Follow-up. Neuromodulation. 2006 Apr;9(2):163-71. doi: 10.1111/j.1525-1403.2006.00056.

ELIGIBILITY:
Inclusion Criteria:

* Refractory overactive bladder syndrome that have an Urgent-SQ tibial nerve implant in 2003-2004

Exclusion Criteria:

* Patient who had the implant removed before the first year after implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory overactive bladder syndrome that have an Urgent-SQ tibial nerve implant
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dick Janssen, MD, Principal Investigator — Radboud University Nijmegen Medical Centre Dept of Urology
Locations (1):
- Radboud Unviversity Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van der Pal F, van Balken MR, Heesakkers JP, Debruyne FM, Bemelmans BL. Implant-Driven Tibial Nerve Stimulation in the Treatment of Refractory Overactive Bladder Syndrome: 12-Month Follow-up. Neuromodulation. 2006 Apr;9(2):163-71. doi: 10.1111/j.1525-1403.2006.00056.x. PMID 22151641